CLINICAL TRIAL: NCT01087177
Title: Evaluating Online Clinical Office-Systems Training to Address SHS Exposure of Children
Brief Title: Effectiveness of Pedialink CEASE Module
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Principal Investigator, Jonathan P. Winickoff, MD, MPH, Associate Professor in Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2007p-001734
Record Dates: First submitted 2010-03-12; First posted 2010-03-16 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Tobacco Use
Keywords: Smoking; Tobacco; Pediatrics
MeSH Terms: conditions — Tobacco Use; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exposure to Pedialink CEASE Trained Site (Experimental): Parents at a practice where the clinicians were trained to address tobacco use through the Pedialink CEASE module.
  Interventions: Other: Exposure to practice that has been trained in Pedialink CEASE

INTERVENTIONS:
Other: Exposure to practice that has been trained in Pedialink CEASE — Child has had an appointment at a practice that was trained in Pedialink CEASE at the time of the interview.

SUMMARY:
The study involves the testing of a Pedialink module through parent exit interviews in one intervention practice and one control practice. Pedialink is the American Academy of Pediatrics' online home for continuous professional development. The intervention site will complete the Pedialink module and the control site will be given routine tobacco control materials.

We will measure changes in practice patterns in the two pediatric practices following the implementation of the online training. At each of these practices, the parents or guardians of children seen by the practice will be surveyed for a one week period before, and a one week period six weeks after either using the online training module (intervention) or being given routine tobacco materials (control).

A follow-up telephone survey will be given to some parents at 3-months. Those given the telephone survey are parents or guardians who smoke or parents or guardians who live with a smoker and are surveyed at the second time-point.

We hypothesize that intervention practices will have higher rates of screening for home and car no-smoking rules and higher rates of advising for home and car no-smoking rules.

DETAILED DESCRIPTION:
This study will involve developing an online training and dissemination system to train pediatricians to address the secondhand smoke exposure of children. We will gather pediatric staff responses to the specific components of the online training and refine this training for a range of outpatient pediatric office settings. We will test the feasibility and efficacy of implementing the online training and dissemination system within the pediatric office setting. We will also gather parental responses to specific components of the pediatric visit, which will be impacted by the online training for pediatric offices.

The following hypotheses will be tested:

Primary Hypothesis

H1. The following measures of physician behavior, as assessed by exit interviews, 3 month follow up telephone interviews of parents or guardians who smoke or parents or guardians who live with a smoker and chart review of 20 charts, will increase more in the intervention practice than in the control practice:

* Screening for home no-smoking rule
* Screening for car no-smoking rule
* Advising parents about the need for a strictly enforced no-smoking in the home rule
* Advising parents about the need for a strictly enforced no-smoking in the car rule.

Secondary Hypothesis H2. Compared to the control practice, the intervention practice will have a greater increase in the summary scores that measure the key processes of practice implementation shown to predict successful practice change. This implementation process will be measured by administering previously validated surveys to physicians and key practice staff before and following the implementation of the office system.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian of child seen by the practice.
* Smoke or live with a smoker.
* Speak English or Spanish.

Exclusion Criteria:

* Under 18
* Cannot be reached by telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Rate of home and car no smoking rules. | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Winickoff, MD, MPH, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hipple B, Nabi-Burza E, Hall N, Regan S, Winickoff JP. Distance-based training in two community health centers to address tobacco smoke exposure of children. BMC Pediatr. 2013 Apr 17;13:56. doi: 10.1186/1471-2431-13-56. PMID 23594832
- See also: CEASE Website — http://www.ceasetobacco.org